CLINICAL TRIAL: NCT04864028
Title: Energy Adaptations During Active Workstation Use: Strategy for Individualization of Active Desk Programs
Brief Title: Energy Profile and Low Intensity Activity (PROFILE)
Acronym: PROFILE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Laboratory AME2P UR3533 (Unknown); Université d'Auvergne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RBHP 2020 DUCLOS 3; 2020-A03311-38 (Other: ANSM)
Record Dates: First submitted 2021-04-09; First posted 2021-04-28 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Healthy
Keywords: Active workstation; cycling; energy expenditure; sedentary
MeSH Terms: conditions — Sedentary Behavior | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volunteer (Experimental)
  Interventions: Other: physical activity

INTERVENTIONS:
Other: physical activity — 15min sitting, 15min standing, 15min sitting, 15 min low intensity cycling

SUMMARY:
The recent literature has highlighting the importance of the time of SB and the level of physical activity (PA) as predictors of metabolic cardio risks. Now, sedentary lifestyles are well recognized as one of the causes of mortality. As with physical activity, a dose-response relationship appears to exist: mortality would increase with time spent in sedentary behaviors. However, this relationship would not be linear: the more the daily sitting time increases, the more the consequences on mortality are important. It is now well demonstrated that time spent in sedentary adult behaviour finds primarily its origin in the work, characterized by prolonged and uninterrupted periods of sitting. Many strategies have been settled to break the prolonged sitting time. The most promising one seem to be the use of active workstations (standing, walking, cycling, stepping) because they reduce sedentary time at work and increase physical activity with positive effects on the global health. However inter variability in energy response have been identified during a sit to stand allocation with subject "savers" profile showing an increase in energy expenditure while others categorized as "non-savers" increased significantly their energy expenditure between sitting and standing position. As others active workstation strategies exist, this study aim to first, better characterize energy response to posture and activity allocation (15min sit-15min stand-15min sit-15min low intensity cycling), secondly to identify parameters that could explain different energy profile.

DETAILED DESCRIPTION:
Subject will have an inclusion visit during a medical consultation where the eligibility criteria to participate to this study will be checked.

During a second experimental visit, subjects will have to take a calibrated breakfast. Three hours after the breakfast, body composition will be assessed and energy expenditure and substrates oxidation will be measured with an indirect calorimetry device during 15min in a sitting position fallowed by 15min in standing position , 15min in a sitting position and 15min of low intensity cycling with a cycling desk.

Then subjects will underwent physical capacity test :

* 6min step test
* Handgrip test
* lower limb strength test Finally, subjects will be equipped with accelerometer and inclinometer device they will need to wore during 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer, male or female, between 18 and 61 years old
* Body mass index > 18,5 kg/m2 and ≤ 25 kg/m2
* Able to provide informed consent to research participation
* Registered in the French social security system

Exclusion Criteria:

* Subject using a sit-to-stand office desk or a swiss ball
* Contact jobs (face-to-face with people)
* Pregnant or breastfeeding women
* Medical or surgical history determined by principal investigator to be not compatible with the study
* Subject with cardiorespiratory and/or osteo-articular disorders limiting their ability to perform physical tests or the use of active offices
* Subject with type 1 or type 2 diabetes treated with insulin
* Subject with progressive cardiovascular or neoplastic disease.
* Subject with a major infection within 3 months of inclusion.
* Subject with known neuromuscular pathology: myopathy, myasthenia, rhabdomyolysis, paraplegia, hemiplegia
* Subject with chronic or acute inflammatory pathology 3 months prior to inclusion

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2023-06-29 (Actual)

PRIMARY OUTCOMES:
energy expenditure | change from baseline to the experimental visit (Day 1)
  Using an indirect calorimetry device change in energy expenditure will be assed during the 1h posture /activity allocation (15min sitting, 15min standing, 15min sitting, 15 min low intensity cycling)

SECONDARY OUTCOMES:
physical activity level (ActiGraph) | during the 7 days following the experimental session
  using acceleometry device (ActiGraph Gt3x)
physical activity level (ActivPAL) | during the 7 days following the experimental session
  using accelerometry (ActivPAL)
Body composition : fat mass and fat free mass | day 0
  body composition will be assessed by bioelectrical impedance device (TANITA MC-780MA)
upper limb strength | during the experimental session after energy expenditure assessment (Day 1)
  will be assessed with handgrip for upper limb muscle
aerobic fitness | during the experimental session after energy expenditure assessment (day 1)
  will be assessed with the Step Test 6 minutes
lower limb strength | during the experimental session after energy expenditure assessment (day1)
  will be assessed with isokinetic dynamometer
eating profile with DEBQ questionnaire (Dutch Eating Behavior Questionnaire) | during the experimental session before energy expenditure assessment (day 1)
  the questionnaire will identify with a scale (items to rank between never and always) three major factors influencing eating behavior "emotional , restrained and external eating". For all items score goes from 0 to 5pts and the lower score the better/healthier.
eating profile with TFEQ questionnaire (Three-Factor Eating Questionnaire) | during the experimental session before energy expenditure assessment (day 1)
  the questionnaire will identify with a scale (items to rank between never and always) three major eating profiles (cognitive restraint, disinhibition, hunger). For Items 1 to 16 score goes from 4 to 1pts, from items 17-21 score goes from 1 to 4 pts. Global score is calculated the lower the healthier.

CONTACTS AND LOCATIONS:
Overall Officials: Martine Duclos, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France